CLINICAL TRIAL: NCT04572295
Title: An Open-label Phase 1b Study of E7090 Monotherapy and in Combination With Other Anticancer Agents in Subjects With ER+, HER2- Recurrent/Metastatic Breast Cancer
Brief Title: A Study of E7090 as Monotherapy and in Combination With Other Anticancer Agents in Participants With Estrogen Receptor Positive (ER+) and Human Epidermal Growth Receptor 2 Negative (HER2-) Recurrent/Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7090-J081-102
Record Dates: First submitted 2020-09-30; First posted 2020-10-01 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-03

CONDITIONS: Breast Neoplasms
Keywords: E7090; Fulvestrant; Exemestane; Receptors, Fibroblast Growth Factor
MeSH Terms: conditions — Breast Neoplasms; Acrocephalosyndactylia | interventions — Fulvestrant; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 Dose Escalation: E7090 + Fulvestrant or Exemestane (Experimental): Participants will receive E7090 tablets, orally, once daily along with fulvestrant 500 milligram (mg), intramuscular injection on Days 1 and 15 of Cycle 1 and each Day 1 of cycle 2 or later, or along with exemestane 25 mg tablet, orally, once daily in 28 days cycle. Each cycle length equals to (=) 28 days.
  Interventions: Drug: E7090; Drug: Fulvestrant; Drug: Exemestane
- Part 2 Monotherapy: E7090 (Experimental): Participants will receive E7090 tablets, orally, once daily in 28 days cycle. Each cycle length =28 days.
  Interventions: Drug: E7090
- Part 3 Dose Expansion: E7090 + Fulvestrant (Experimental): Participants will receive E7090 tablets, orally, once daily along with fulvestrant 500 mg, intramuscular injection on Days 1 and 15 of Cycle 1 and each Day 1 of cycle 2 or later. Each cycle length =28 days.
  The dose of E7090 for Part 3 in combination with fulvestrant will be determined based on the safety, tolerability, pharmacokinetic (PK), and biomarker data obtained from Part 1.
  Interventions: Drug: E7090; Drug: Fulvestrant

INTERVENTIONS:
Drug: E7090 — E7090 oral tablet.
Drug: Fulvestrant — Fulvestrant intramuscular injection.
  Arms: Part 1 Dose Escalation: E7090 + Fulvestrant or Exemestane; Part 3 Dose Expansion: E7090 + Fulvestrant
Drug: Exemestane — Exemestane oral tablet.
  Arms: Part 1 Dose Escalation: E7090 + Fulvestrant or Exemestane

SUMMARY:
The primary purpose of this study is to evaluate the tolerability and safety of E7090 as monotherapy and in combination with other anticancer agents in participants with ER+, HER2- recurrent/metastatic breast cancer and to determine the recommended dose (RD) of E7090 in combination with other anticancer agents for subsequent phase studies.

ELIGIBILITY:
Inclusion Criteria:

Common to Part 1, 2 and 3

1. Participants who provided written voluntary informed consent for participation in the study.
2. Female participants who are age >=18 years at the time of informed consent.
3. Post-menopausal or pre/peri-menopausal participants who have been continuously on concurrently given a luteinizing hormone-releasing hormone (LHRH) agonist since before the start of study treatment and is planned to continue this treatment during the study.
4. Participants with histologically confirmed diagnosis of progressive/recurrent or metastatic, ER+, HER2 negative breast cancer.
5. Participants who received prior CDK4/6 inhibitor treatment.
6. Participants with Performance Status (PS) score of 0-1 established by Eastern Cooperative Oncology Group (ECOG).
7. Part 1 and Part 2: Participants with at least one accessible lesion for biopsy and who agree to undergo a biopsy of accessible lesion prior to study treatment (if archived tissues collected after CDK4/6 inhibitor treatment is not available) and on Day 1 of Cycle 3.

   (Part 3) participants must agree to undergo a biopsy at screening if no archival tissue is available (tissue collection must be after CDK4/6 inhibitor treatment and prior to study treatment). A biopsy on Day 1 of Cycle 3 is not mandatory.
8. Participants who agree to provide archival or fresh tumor tissue collected after CDK4/6 inhibitor treatment.
9. Part 2 only: Participants with positive protein expression of fibroblast growth factor receptor 1 (FGFR) and/or FGFR2, with which tumor was collected after CDK4/6 inhibitor treatment at the central laboratory.

Exclusion criteria:

1. Participants with brain or subdural metastases, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment in this study. Any signs (example. radiologic) or symptoms of brain metastases must be stable for at least 4 weeks before starting study treatment.
2. (Part 1 and Part 2) Participant who have received 2 or more regimen of chemotherapy for the treatment of advanced or metastatic lesions.
3. (Part 3) Participant who have received 1 or more regimens of chemotherapy or antibody-drug conjugate therapy for the treatment of advanced or metastatic lesions.
4. Participant with inflammatory breast cancer.
5. Participant with bilateral breast cancer of different histologic types. Participants who have bilateral breast cancers that are both ER+ and HER2- may be enrolled in the study.
6. Participant who have history of active malignancy within the past 24 months prior to the first dose of study drugs.
7. Participants with clinically significant cardiovascular impairment.
8. Presence of a progressive central nervous system (CNS) disease, including degenerative CNS diseases and progressive tumors.
9. Concomitant active infection requiring systemic treatment.
10. Participants who test positive for human immunodeficiency virus (HIV antibody), or positive for hepatitis B surface (HBs antigen) or hepatitis C (HCV antibody and RNA).
11. Participants with following ocular disorders:

    1. Current evidence of Grade 2 or higher corneal disorder.
    2. Current evidence of active retinopathy (example. age-related macular degeneration, central serous chorioretinal disease, retinal tear)
12. Participants who received prior treatment with an FGFR inhibitor.
13. Females who are pregnant or breastfeeding.
14. Part 1 only: Participants with T-score less than (<) -2.5 by dual-energy X-ray absorptiometry (DXA) scan.
15. Part 3 only: Participants who received 3 or more prior lines of endocrine therapy in advanced/metastatic setting.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 51 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Recommended Dose (RD) of E7090 in Combination With Other Anticancer Agents | Up to Cycle 1 (each cycle length = 28 days)
Part 1: Number of Participants With Dose-limiting Toxicities (DLTs) | Up to Cycle 1 (each cycle length = 28 days)
  DLTs will be assessed based on combination regimen-related adverse events (AEs) occurred during Cycle 1 of Part 1 and the severity of AEs will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 30 days after last administration of study drug (approximately up to 66 months)
  Safety assessments will consist of monitoring and recording all AEs and SAEs; regular measurement of vital signs and ECG; and regular monitoring of clinical laboratory parameters, body weight and bone density.

SECONDARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration of E7090, its Metabolite (M2) and Exemestane | For E7090 and its metabolite (M2)- Parts 1 and 2 Cycle 1 Day 1: 0-24 hours post-dose; For exemestane- Part 1 Cycle 1 Day 1: 0-24 hours post-dose (each cycle length = 28 days)
AUC: Area Under the Plasma Concentration-time Curve of E7090, its Metabolite (M2) and Exemestane | For E7090 and its metabolite (M2)- Parts 1 and 2 Cycle 1 Day 1: 0-24 hours post-dose; For exemestane- Part 1 Cycle 1 Day 1: 0-24 hours post-dose (each cycle length = 28 days)
Part 1: Plasma Concentration of Fulvestrant | Cycles 2 and 3 Day 1: pre-dose (each cycle length = 28 days)
Objective Response Rate (ORR) | Baseline up to 66 months
  The ORR will be assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. ORR is defined as a percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR). CR: disappearance of all lesions. PR: For PR, longest diameter will be used for non-lymph target lesions but short axis is measured for lymph lesions. PR: greater than or equal to (>=) 30 percent (%) decrease in sum of diameters of target lesions taking as reference baseline, associated to non-progressive disease (non-PD) response for non-target (NT) lesions.
Disease Control Rate (DCR) | Baseline up to 66 months
  DCR will be assessed according to RECIST version 1.1. DCR is defined as a percentage of participants with BOR of CR, PR or stable disease (SD). The BOR of SD has to be observed >=7 weeks from the date of first study dose. CR: disappearance of all lesions. PR: For PR, longest diameter will be used for non-lymph target lesions but short axis is measured for lymph lesions. PR: >=30% decrease in sum of diameters of target lesions taking as reference baseline, associated to non-PD response for NT lesions.
Clinical Benefit Response (CBR) | Baseline up to 66 months
  CBR will be assessed according to RECIST version 1.1. CBR is defined as a percentage of participants with BOR of CR, PR or durable SD (dSD) (duration of SD >=23 weeks). CR: disappearance of all lesions. PR: For PR, longest diameter will be used for non-lymph target lesions but short axis is measured for lymph lesions. PR: >=30% decrease in sum of diameters of target lesions taking as reference baseline, associated to non-PD response for NT lesions.
Progression-free Survival (PFS) | Baseline up to 66 months
  PFS will be assessed according to RECIST version 1.1. PFS is defined as the time from the date of first dose to the date of first documentation of disease progression or date of death from any cause, whichever occurs first.
Overall Survival (OS) | Baseline up to 66 months
  OS is defined as the time from the date of first dose to the date of death from any cause.
Time to Response (TTR) | Baseline up to 66 months
  TTR will be assessed according to RECIST version 1.1. TTR is defined as the time from the date of first study dose to the date of first documentation of CR or PR. CR: disappearance of all lesions. PR: For PR, longest diameter will be used for non-lymph target lesions but short axis is measured for lymph lesions. PR: >=30% decrease in sum of diameters of target lesions taking as reference baseline, associated to non-PD response for NT lesions.
Duration of Response (DOR) | Baseline up to 66 months
  DOR will be assessed according to RECIST version 1.1. DOR is defined as the time from the date of first documentation of CR or PR to the date of first documentation of disease progression or date of death from any cause, whichever occurs first. CR: disappearance of all lesions. PR: For PR, longest diameter will be used for non-lymph target lesions but short axis is measured for lymph lesions. PR: >=30% decrease in sum of diameters of target lesions taking as reference baseline, associated to non-PD response for NT lesions.

CONTACTS AND LOCATIONS:
Locations (11):
- Japan (11):
  - Eisai Trial Site 11, Nagoya, Aichi-ken
  - Eisai Trial Site 6, Kashiwa, Chiba
  - Eisai Trial Site 9, Matsuyama, Ehime
  - Eisai Trial Site 5, Yokohama, Kanagawa
  - Eisai Trial Site 4, Sendai, Miyagi
  - Eisai Trial Site 7, Chuo-ku, Osaka
  - Eisai Trial Site 10, Kitaadachi-gun, Saitama
  - Eisai Trial Site 3, Chuo-ku, Tokyo
  - Eisai Trial Site 1, Koto-ku, Tokyo
  - Eisai Trial Site 2, Shinagawa-ku, Tokyo
  - Eisai Trial Site 8, Shinjuku-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.